CLINICAL TRIAL: NCT01197781
Title: An Open-label, Single-Centre Study to Assess the Pharmacokinetics of R406 in Healthy Volunteers When Fostamatinib Disodium 150 mg is Administered Alone and in Combination With Verapamil
Brief Title: Evaluation of the Drug-drug Interaction Between FosD and Verapamil When Taken Together in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00011
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Drug Drug Interactions; Healthy Volunteers
Keywords: Phase I; FosD; fostamatinib disodium; verapamil; healthy volunteers
MeSH Terms: interventions — Verapamil

ARMS (2):
- Period 1 (Experimental)
  Interventions: Drug: FOSTAMATIN
- Period 2 (Experimental)
  Interventions: Drug: FOSTAMATIN; Drug: Verapamil

INTERVENTIONS:
Drug: FOSTAMATIN — Oral tablets - single dose
Drug: Verapamil — Oral tablets - administered 3 times daily over 4 days
  Arms: Period 2

SUMMARY:
This Study evaluates the possible drug interaction between FosD and verapamil when taken together.

DETAILED DESCRIPTION:
An Open-label, Single-Centre Study to Assess the Pharmacokinetics of R406 in Healthy Volunteers when Fostamatinib Disodium 150 mg is Administered Alone and in Combination with Verapamil.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 50 kg (110 lbs) and body mass index (BMI) between 18 and 35 kg/m2, inclusive.
* Females must be of non-childbearing potential

Exclusion Criteria:

* History of clinically significant disease or disorder or presence of GI, hepatic or renal disease
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the drug
* Any clinically significant abnormalities in lab safety tests or vital signs as results as judged by the Investigator
* Use of prescription or over-the-counter drugs within 2 weeks of first administration of investigational product
* Current smokers or use of nicotine products within 1 month prior to enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine plasma PK parameters of R406 when FosD is given in combination with verapamil (including but not limited to: AUC, tmax, Cmax and terminal elimination half life (t1/2)) of FosD. | Daily during Treatment Period 1 (FosD alone) and Treatment Period 2 (FosD plus verapamil) until 96 hours post each single dose of FosD

SECONDARY OUTCOMES:
To investigate safety and tolerability of FosD when given in combination with verapamil: adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, ECGs. | Screening, throughout both treatment periods, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca; Carlos Prendes, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Recruiting Site, Overland Park, Kansas, United States